CLINICAL TRIAL: NCT01347346
Title: Phase I/II Clinical Trial of Haematopoietic Stem Cell Gene Therapy for the Wiskott-Aldrich Syndrome
Brief Title: Gene Therapy for WAS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genethon (Other)
Collaborators: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTG003.08; 2009-011152-22 (EudraCT Number)
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Wiskott-Aldrich Syndrome
Keywords: Wiskott-Aldrich Syndrome; Primary immune deficiency; ex vivo gene therapy; hematopoietic stem cells
MeSH Terms: conditions — Wiskott-Aldrich Syndrome; Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: Autologous CD34 positive cells transduced with a lentiviral vector containing human WAS gene — transplantation of patient's autologous CD34+ cells transduced with lentiviral vector containing human WAS gene

SUMMARY:
This is a phase I/II study to evaluate the safety and efficacy of Hematopoietic Stem Cell genetherapy for the Wiskott-Aldrich Syndrome.

DETAILED DESCRIPTION:
This clinical trial is an ex vivo gene therapy trial. The investigational product corresponds to autologous CD34+ cells transduced with a lentiviral vector harboring the human WASP gene.

ELIGIBILITY:
Inclusion Criteria:

* males of all ages
* severe WAS (clinical score 3-5) or absence of WAS protein in peripheral blood mononuclear cells determined by Western blotting and flow cytometry
* molecular confirmation by WAS gene DNA sequencing
* lack of HLA-genotypically identical bone marrow after 3 month search
* lack of a 10/10 or 9/10 antigen HLA-matched unrelated donor after 3 month search
* lack of a HLA-matched cord blood after 3 month search
* parental, guardian, patient signed informed consent/assent
* willing to return for follow-up
* only for patients who have received previous allogenic hematopoietic stem cell transplant:
* failed allogenic hematopoietic stem cell transplant
* contraindication to repeat transplantation

Exclusion Criteria:

* patient with HLA-genotypically identical bone marrow
* patient with 10/10 or 9/10 antigen HLA-matched unrelated donor or with HLA-matched cord blood
* contraindication to leukapheresis
* contraindication to bone marrow harvest
* contraindication to administration of conditioning medication
* HIV positive patient

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2016-01-13 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Improvement in the eczema status | 2 years
  Improvement in eczema status as compared with the baseline status at study entry on clinical evaluation
Reduction in the frequency and severity of infection episodes | 2 years
  Reduction in the frequency and severity of infection episodes as compared with the baseline status and the patient's historical data collected over the 2 years prior to study entry
Reduction in the frequency and severity of bruising and bleeding episodes | 2 years
  Reduction in the frequency and severity of bruising and bleeding episodes as compared with the baseline status and the patient's historical data collected over the 2 years prior to study entry
Reduction in the frequency and severity of autoimmune disorders | 2 years
  Reduction in the frequency and severity of autoimmune disorders as compared with the baseline status at study entry
Reduction in the number of disease related days of hospitalization | 2 years
  Reduction in the number of disease related days of hospitalization as compared with the patient's historical data collected over the 2 years prior to study entry

SECONDARY OUTCOMES:
Occurrence and type of adverse events | 2 years
  Occurrence and type of adverse events reported during the course of the study
Change in medical conditions | 2 years
  Assessment of weight, vital signs, ECG and laboratory exams during the course of the study
Safety of lentivirus gene transfer into Hematopoietic Stem Cells | 3, 6, 12, 24 months / 6, 12, 18, 24 months
  Detection of replication competent lentivirus (RCL) and lentivirus integration sites analysis
Improvement of microthrombocytopenia | 3, 6, 12, 24 months
  Improvement of microthrombocytopenia as compared with the baseline evaluation at study entry
Decrease in the number and volume of platelets transfusions | 2 years
  Decrease in the number and volume of platelets transfusions as compared with patient's historical data collected over the 2 years prior to study entry
Evidence of sustained engraftment of WASP-expressing transduced cells | 6 weeks, 1, 3, 6, 9, 12, 18 & 24 months
  Quantification of vector copy numbers and detection of vector-derived WASP expression
Reconstitution of humoral and cell mediated immunity | 9, 12, 18 & 24 months
  Reconstitution of humoral and cell mediated immunity as compared with the baseline evaluation at study entry

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

REFERENCES:
- [Derived] Magnani A, Semeraro M, Adam F, Booth C, Dupre L, Morris EC, Gabrion A, Roudaut C, Borgel D, Toubert A, Clave E, Abdo C, Gorochov G, Petermann R, Guiot M, Miyara M, Moshous D, Magrin E, Denis A, Suarez F, Lagresle C, Roche AM, Everett J, Trinquand A, Guisset M, Bayford JX, Hacein-Bey-Abina S, Kauskot A, Elfeky R, Rivat C, Abbas S, Gaspar HB, Macintyre E, Picard C, Bushman FD, Galy A, Fischer A, Six E, Thrasher AJ, Cavazzana M. Long-term safety and efficacy of lentiviral hematopoietic stem/progenitor cell gene therapy for Wiskott-Aldrich syndrome. Nat Med. 2022 Jan;28(1):71-80. doi: 10.1038/s41591-021-01641-x. Epub 2022 Jan 24. PMID 35075289